CLINICAL TRIAL: NCT06874010
Title: A Phase 1/2, Open-Label, Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Subcutaneous and Intravenous DT-216P2 in Patients With Friedreich's Ataxia
Brief Title: A Multiple Ascending Dose Study of DT-216P2 in Patients With Friedreich's Ataxia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Design Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DTX-216P2-101
Record Dates: First submitted 2025-02-25; First posted 2025-03-13 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DT-216P2 (Experimental)
  Interventions: Drug: DT-216P2

INTERVENTIONS:
Drug: DT-216P2 — Active

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, and pharmacokinetics of DT-216P2 administered multiple ascending doses in patients with FA.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18-65 years of age inclusive, at the time of signing the informed consent.
* Genetically confirmed diagnosis of FA, with homozygous GAA repeat expansions in the frataxin gene.
* Stage 5.5 or less on the FSA at screening.
* BMI between 16 and 32 kg/m2 at screening; weight should be <= 100 kg at screening.
* Male and/or female using protocol defined and regulatory approved contraception.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Any concomitant medical condition that in the opinion of the investigator, puts the participant at risk or precludes participant from completing the study protocol.
* Any clinically significant nonmedical conditions and psychiatric disorders that could put the participant at higher risk for participation in the study, influence the participant's ability to participate in the study, or interfere with interpretation of the participant's study results, in the opinion of the investigator.
* Received an investigational agent within the last 30 days or 5 half-lives, whichever longer, prior to the first dose of study drug, or are in follow-up of another clinical study prior to study enrollment. Exception: Potential participants who are currently on Omaveloxolone must be on stable doses for at least 3 months.
* Is not willing to comply with the contraceptive requirements during the study period, as per protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events (TEAE) | Up to Week 12

SECONDARY OUTCOMES:
Area under the curve (AUClast, AUCinf) | Up to Week 12
Maximum concentration (Cmax) | Up to Week 12
Time to Cmax (Tmax) | Up to Week 12
Half-life (t1/2) | Up to Week 12
Frataxin expression at baseline and after treatment will be measured | Up to Week 12

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Scientia Clinical Research Ltd, Sydney, New South Wales
  - Doherty Clinical Trials, East Melbourne, Victoria
  - Nucleus Network, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No